CLINICAL TRIAL: NCT05646043
Title: PREHABILITATION During Neoadjuvant Therapy in Patients With Cancer of the Upper Digestive Tract and Rectum
Brief Title: PREHAB - Improving Condition Before Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 08/RVO-FNOs/2022
Record Dates: First submitted 2022-11-15; First posted 2022-12-12 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Cancer, Digestive System; Cancer, Rectum
Keywords: prehabilitation; cancer of the digestive system; cancer of the rectum; endurance walking; power training
MeSH Terms: conditions — Digestive System Neoplasms; Rectal Neoplasms | interventions — Physical Conditioning, Human

STUDY DESIGN:
Intervention Model Description: The study subjects will be enrolled in two parallel groups.
Masking Description: No masking is used in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with cancer of the digestive system (Active Comparator): Patients with cancer of the digestive system (oesophageal and stomach cancer) will be enrolled in this study arm.
  Interventions: Behavioral: Physical training; Behavioral: Muscle strength training
- Patients with cancer of the rectum (Active Comparator): Patients with cancer of the rectum will be enrolled in this study arm.
  Interventions: Behavioral: Physical training; Behavioral: Muscle strength training

INTERVENTIONS:
Behavioral: Physical training — Physical training consists of endurance walking and strength training. The basis for determining the number of steps per day is the baseline value of each patient. This will increase by 10-15% every week until the surgery date. The assumption of a total load increase is 120-180% compared to the baseline.
Behavioral: Muscle strength training — Muscle strength training will take place using exercises to strengthen the upper and lower limbs and to strengthen the trunk. There will be a set of 5 exercises in two difficulty variants. The study subjects will perform this set 7 days a week, and will repeat the assembly a total of two times. The total time of strength training is 10 min.

SUMMARY:
The pilot research project is focused on the feasibility of a prehabilitation program for two groups of diagnoses (esophageal and stomach cancer, rectal cancer).

DETAILED DESCRIPTION:
With the aim of achieving downstaging, downsizing, and reducing the risk of recurrence, neoadjuvant chemotherapy, possibly chemoradiotherapy - i.e. neoadjuvant therapy is indicated in the preoperative period for patients with cancer of the upper digestive tract and rectal cancer.

Chemotherapy has a negative impact not only on the overall physical and mental condition of the patient but also on the quality of life and on the daily activities of the individual, especially in the period when the organism is facing an abnormal stress load in the sense of extensive surgical procedures.

Recently, attention and efforts to improve postoperative morbidity and mortality have increasingly focused on the preoperative period. The concept of prehabilitation, which is defined as an intervention improving functional capacity before an upcoming physiological stressor, appears as a way to contribute to this. This fact is evidenced by a number of published references.

The main aim of the study is to confirm or refute the feasibility of the prehabilitation program during neoadjuvant therapy in two diagnostic groups of patients:

* - Patients with cancer of the upper digestive tract
* - Patients with rectal cancer

The prehabilitation program will be implemented in the patient's home environment.

The study aims to answer the basic research question of whether selected patients will be able to complete a home exercise regimen during the preoperative period when they will undergo neoadjuvant therapy.

As part of the study, the program's security and feasibility will be tested.

ELIGIBILITY:
Inclusion Criteria:

* radically operable locally advanced cancer of the esophagus, esophagogastric junction, stomach
* radically operable locally advanced carcinoma of the rectum
* the patient is able to handle the planned surgical resection procedure
* planned preoperative neoadjuvant therapy
* age > 18 years
* the ability to complete a spiroergometric examination
* the ability to carry out a prehabilitation program consent to participate in the study confirmed by signing the informed consent

Exclusion Criteria:

* contraindications for spiroergometric examination
* limitation on the part of the locomotor system to spiroergometric examination or daily exercise (e.g. amputation, severe gonarthrosis, coxarthrosis)
* inoperability determined by the interdisciplinary team
* inability to manage the planned operational performance
* acute surgical performance
* synchronous malignant disease
* multivisceral resection
* planned non-surgical therapeutic procedure
* incomplete data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of enrolled patients | 3 months
  The number of patients who express an interest in being included in the study from all patients diagnosed and indicated for neoadjuvant therapy in the monitored period. the reasons for refusal to enroll in the study will be monitored.
Number of patients completing the program | 3 months
  The number of patients who complete the prehabilitation program by the time of surgery.
Individual patient compliance | 3 months
  Number of days when the patient wore the smart bracelet and performed or attempted to perform the exercise program out of the total number of days in the monitored period

SECONDARY OUTCOMES:
Changes in spirometry examination results | 3 months
  Changes in spirometry examination will be assessed, comparing the baseline values with the values after training (maximum tidal volume (ml/1kg of weight/1 min), anaerobic threshold (beats/min).
Changes in the quality of life | 3 months
  Changes in the quality of life will be monitored using the EORTC Core Quality of Life questionnaire (EORTC QLQ-C30). This questionnaire is designed to measure cancer patients' physical, psychological and social functions.
Parameters monitored by the oncologist | 3 months
  Number of patients with chemotherapy dose reduction or premature termination of chemotherapy, number of patients with complete chemotherapy, number of patients hospitalized due to chemotherapy toxicity
Exercise program - number of steps/day | 3 months
  The number of steps taken by the study subjects in a day will be counted.
Exercise program - pressing force on the dynamometer | 3 months
  The pressing force on the dynamometer (in kg) will be assessed at the beginning and at the end of the program.
Exercise program - InBody examination | 3 months
  The InBody examination (analysis of body composition in %) will be performed at the beginning and at the end of the program.
Exercise program - Body Mass Index | 3 months
  The value of Body Mass Index will be recorded at the beginning and at the end of the program will be assessed (in kg/m2), changes will be assessed.
Exercise program - perceived exertion | 3 months
  The perceived exertion will be assessed using the Borg Rating of Perceived Exertion Scale (RPE). RPE is based on the physical sensations a person experiences during physical activity, including increased heart rate, increased respiration or breathing rate, increased sweating, and muscle fatigue. The rating is from 6 to 20.
Parameters monitored by the anesthesiologist - ASA value | 3 months
  ASA value - the ASA physical status classification system is a system for assessing the fitness of patients before surgery. It is a five-category physical status classification defined by the American Society of Anesthesiologists.
Parameters monitored by the anesthesiologist - morbidity assessment | 3 months
  Morbidity assessment among the study population will be performed, using assessment of incidence and prevalence.
Parameters monitored by the anesthesiologist - preoperative analgesia | 3 months
  The use of preoperative analgesia will be recorded and assessed.
Parameters monitored by the anesthesiologist - postoperative opioid analgesia | 3 months
  The use of postoperative opioid analgesia will be recorded and assessed.
Parameters monitored by the anesthesiologist - pain assessment | 3 months
  The Numeric Pain Rating Scale will be used to assess pain. The Numeric Pain Rating Scale is a unidimensional measure of pain intensity in adults, including those with chronic pain due to rheumatic diseases.
Laboratory examinations - complete blood count | 3 months
  Complete blood count will be analyzed (g/L).
Laboratory examinations - CRP values | 3 months
  C-Reactive Protein (CRP) will be assessed (in mg/L). C-reactive protein (CRP) is an acute phase protein that is produced in the liver. The levels increase rapidly in response to acute inflammation.
Laboratory examinations - procalcitonin level | 3 months
  Procalcitonin levels will be analyzed (ng/L). This marker indicates the presence of infection.
Laboratory examinations - nutritional parameters | 3 months
  Nutritional parameters - the levels of total protein, albumin and prealbumin will be analyzed (mg/dL).
Laboratory examinations - coagulation factors (aPTTp | 3 months
  Coagulation factors - Activated Partial Thromboplastin Time (APTT) will be measured (in seconds).
Laboratory examinations - coagulation factors (fibrinogen) | 3 months
  Coagulation factors - fibrinogen levels will be assessed (mg/dL). Higher and lower levels point to blood clotting disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Irina Chmelová, MD,PhD,MBA, Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers. The data may be provided upon request.

REFERENCES:
- [Derived] Chmelova I, Pastucha D, Hudecek T, Guran Z, Ciecotkova S, Martinek L, Zubikova J, Matlova A, Dolezel J, Salounova D, Chmelo J. Prehabilitation during neoadjuvant therapy in patients with cancer of the upper gastrointestinal tract and rectum-the study protocol. Front Sports Act Living. 2025 Feb 3;6:1495398. doi: 10.3389/fspor.2024.1495398. eCollection 2024. PMID 39963182